CLINICAL TRIAL: NCT06008808
Title: An Open-Label Phase I Study of JAK Inhibitor Ruxolitinib With and Without CTLA-4 Ig Abatacept for the Prophylaxis of Graft-Versus-Host Disease and Cytokine Release Syndrome After T-cell Replete Haploidentical Peripheral Blood Hematopoietic Cell Transplantation
Brief Title: Ruxolitinib With and Without CTLA-4 Ig Abatacept for the Prophylaxis of Graft-Versus-Host Disease and Cytokine Release Syndrome After T-cell Replete Haploidentical Peripheral Blood Hematopoietic Cell Transplantation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Incyte Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 202401211
Record Dates: First submitted 2023-08-18; First posted 2023-08-24 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Graft Vs Host Disease; Graft-versus-host-disease; Graft Versus Host Disease
Keywords: Haploidentical; GVHD; CRS
MeSH Terms: conditions — Graft vs Host Disease | interventions — ruxolitinib; Abatacept

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Regimen 1: Ruxolitinib (Experimental): -Ruxolitinib at 5 mg twice per day (BID) beginning on Day -3 and continuing until Day 180 followed by a taper (duration of taper depends on dose of ruxolitinib at Day 180). Once a patient's counts have reached ANC ≥ 1.5 K/cumm, hemoglobin ≥ 9.0 g/dL, and platelets ≥ 50 K/cumm, ruxolitinib dosing will escalate to 10 mg BID.
  Interventions: Drug: Ruxolitinib
- Regimen 2: Ruxolitinib + Abatacept (Experimental): * Ruxolitinib at 5 mg twice per day (BID) beginning on Day -3 and continuing until Day 180 followed by a taper (duration of taper depends on dose of ruxolitinib at Day 180). Once a patient's counts have reached ANC ≥ 1.5 K/cumm, hemoglobin ≥ 9.0 g/dL, and platelets ≥ 50 K/cumm, ruxolitinib dosing will escalate to 10 mg BID.
  * In addition, patients will receive abatacept 10 mg/kg IV over 30 minutes on days +5, +14, +28, and +56.
  Interventions: Drug: Ruxolitinib; Drug: Abatacept

INTERVENTIONS:
Drug: Ruxolitinib — Ruxolitinib is provided by Incyte Corporation.
  Other Names: Jakafi
Drug: Abatacept — Abatacept is commercially available.
  Arms: Regimen 2: Ruxolitinib + Abatacept

SUMMARY:
Allogeneic hematopoietic cell transplantation (HCT) is one of the only curative intent therapies available for hematologic malignancies. HLA-matched sibling donors have historically offered the best clinical results but are unavailable for the majority of patients, while most patients do have readily available haploidentical donors. One of the risks of a haploidentical HCT is graft vs. host disease (GVHD), but it is difficult to reduce the incidence of GVHD without compromising the graft vs. leukemia (GVL) effect.

The hypothesis of this study is that JAK inhibition with and without CTLA-4 Ig with haploidentical HCT may mitigate GVHD and cytokine release syndrome while retaining the GVL effect and improving engraftment.

ELIGIBILITY:
Inclusion Criteria:

Patients must meet the following criteria within 30 days prior to Day -3 unless otherwise noted.

* Diagnosis of one of the hematological malignancies listed below:

  * Acute myelogenous leukemia (AML) in complete morphological remission, complete remission with incomplete hematologic recovery, and complete remission with partial hematologic recovery (based on ELN Criteria47).
  * Acute lymphocytic leukemia (ALL) in complete morphological remission (MRD negative by flow cytometry with sensitivity to ≤ 10-4).
  * Myelodysplastic syndrome with ≤ 10% blasts in bone marrow.
  * Non-Hodgkin lymphoma (NHL) or Hodgkin lymphoma (HD) in second or greater complete or partial remission.
  * Myelofibrosis with ≤ 10% blasts in bone marrow. Up to five patients with myelofibrosis will be permitted in Regimen 1 and up to five in Regimen 2.
  * AML in partial response. One patient will be enrolled in Regimen 1 given the prospect of potential benefit.
* Planned treatment is T cell-replete peripheral blood haploidentical donor transplantation.
* Available HLA-haploidentical donor who meets the following criteria:

  * Blood-related family member, including (but not limited to) sibling, offspring, cousin, nephew, or parent. Younger donors should be prioritized.
  * At least 18 years of age.
  * HLA-haploidentical donor/recipient match by at least low-resolution typing per institutional standards.
  * In the investigator's opinion, is in general good health and medically able to tolerate leukapheresis required for harvesting hematopoietic stem cells.
  * No active hepatitis.
  * Negative for HTLV and HIV.
  * Not pregnant.
  * Donor selection will be in compliance with FDA guidelines as provided in 21 CFR 1271 for donor eligibility https://www.fda.gov/downloads/BiologicsBloodVaccines/GuidanceComplianceRegulatoryInformation/Guidances/Tissue/UCM091345.pdf
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
* Adequate organ function as defined below:

  * Total bilirubin ≤ 1.5 x IULN.
  * AST (SGOT) and ALT (SGPT) ≤ 3.0 x IULN.
  * Creatinine ≤ 1.5 x IULN OR creatinine clearance ≥ 45 mL/min/1.73 m2 by Cockcroft-Gault Formula.
  * Oxygen saturation ≥ 90% on room air.
  * LVEF ≥ 40%.
  * FEV1 and FVC ≥ 40% predicted, DLCOc ≥ 40% predicted. If DLCO is < 40%, patients will still be considered eligible if deemed safe after a pulmonary evaluation.
* Able to receive GVHD prophylaxis with tacrolimus, mycophenolate mofetil (if applicable), and cyclophosphamide.
* At least 18 years of age at the time of study consent
* The effects of ruxolitinib and abatacept on the developing human fetus are unknown. Additionally, tacrolimus may increase risk of hypertension, preeclampsia, preterm birth, and low birth weight; and mycophenolate mofetil is considered to be teratogenic. For this reason, women of childbearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control, abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study and for the duration of the study.
* Able to understand and willing to sign an IRB approved written informed consent document (or that of legally authorized representative, if applicable).

Exclusion Criteria:

* Prior allogeneic transplant (regardless of whether donor was related, unrelated, or cord). Prior autologous transplant is not exclusionary.
* Presence of donor specific antibodies (DSA) with Mean Fluorescence Intensity (MFI) of ≥ 4000 as assessed by the single antigen bead assay.
* Known HIV or active hepatitis B or C infection. Known current history of active tuberculosis.
* Known hypersensitivity to one or more of the study agents.
* Planning to receive antithymocyte globulin as part of the pre-transplant conditioning regimen.
* Currently receiving or has received any investigational drugs within the 14 days prior to the first dose of study drug (Day -3).
* Pregnant and/or breastfeeding. Women of childbearing potential must have a negative pregnancy test within 14 days of Day -3.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, autoimmune disease, symptomatic congestive heart failure, unstable angina pectoris, or unstable cardiac arrhythmias.
* Immunosuppressive doses of steroids. Subjects with steroids for adrenal insufficiency will not be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2026-09-09 (Estimated); Study Completion 2026-12-11 (Estimated)

PRIMARY OUTCOMES:
Cumulative incidence of graft failure | Day 35
Cumulative incidence of grades III-IV acute GVHD by MAGIC criteria | Day 100
Number of patients who experience CRS | Through day 14

SECONDARY OUTCOMES:
Cumulative incidence of grades II-IV acute GVHD by MAGIC criteria | Day 100
Non-relapse mortality | Day 180
  Defined as death from any cause other than disease relapse.
Feasibility of regimen | From day -3 to day 30
  Defined as at least 80% of patients successfully taking at least 80% of the ruxolitinib dose

CONTACTS AND LOCATIONS:
Overall Officials: Ramzi Abboud, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu